CLINICAL TRIAL: NCT02484625
Title: The Effect of Solid, Semi-Solid and Fluid Dairy Products on Short-Term Food Intake and Satiety in Children
Brief Title: The Effect of Dairy and Non-Dairy Snacks on Food Intake, Subjective Appetite in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-001; 2016-130 (Other: Mount Saint Vincent University)
Record Dates: First submitted 2015-04-17; First posted 2015-06-29 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Food; Eating; Appetite
Keywords: Snacking; Food Intake; Satiety; Obesity
MeSH Terms: conditions — Obesity | interventions — Cheese; Milk

STUDY DESIGN:
Intervention Model Description: Randomized crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Potato chips (Experimental): Commercial potato chips, 180 kcal
  Interventions: Other: Potato chips
- Greek yogurt (Experimental): Greek yogurt, 180 kcal
  Interventions: Other: Greek yogurt
- Cookies (Experimental): Sandwich-type cookies, 180 kcal
  Interventions: Other: Cookies
- Cheese (Experimental): Mozzarella cheese, 180 kcal
  Interventions: Other: Cheese
- Milk (fluid) (Experimental): Milk, 2% m.f., 180 kcal
  Interventions: Other: Milk

INTERVENTIONS:
Other: Potato chips — Commercially available potato chips, 180 kcal
  Arms: Potato chips
Other: Greek yogurt — Commercially available Greek yogurt, 180 kcal
  Arms: Greek yogurt
Other: Cookies — Commercially available cookies, 180 kcal
  Arms: Cookies
Other: Cheese — Commercially available cheese, 180 kcal
  Arms: Cheese
Other: Milk — Commercially available milk, 180 kcal
  Arms: Milk (fluid)

SUMMARY:
Dairy products have the potential to be healthy snack foods for children and are provided in a variety of food matrices. For instance, milk represents a fluid product, yogurt can be classified as a semi-solid food, and finally, cheese is the example of solid food. This experiment is aimed to examine the effect of dairy products with different food matrices on satiety and food intake in children. Dairy products will be compared with other non-dairy snacks popular among children including cookies and potato chips.

ELIGIBILITY:
Inclusion Criteria:

* Born at full-term within the normal weight range
* 9-14 year old

Exclusion Criteria:

* Food sensitivities or allergies,
* Dietary restrictions,
* Health, learning, emotional or behavioural problems
* Receiving medication

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Food intake (grams and kcal) measured with a test meal | 120 min
  The amount of energy (kcal) consumed ad libitum with the test meal (pizza lunch) two hours later.
Subjective appetite measured with Visual Analogue Scales | 0-120 min
  The subjective assessment of appetite parameters including a desire to eat, fullness, hunger and a prospective food consumption measured with 100 mm Visual Analogue Scales with two opposite statements at each end (e.g., for the hunger scale, 0 mm means not hungry at all, and 100 mm means very hungry).

SECONDARY OUTCOMES:
Cortisol | 0-120 min
  The concentration of salivary cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan L Luhovyy, PhD, Principal Investigator — Mount Saint Vincent University
Locations (1):
- Mount Saint Vincent University, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Gheller BJF, Li AC, Gheller ME, Armstrong T, Vandenboer E, Bellissimo N, Anini Y, Hamilton J, Nunes F, Mollard RC, Anderson GH, Luhovyy BL. The effect of dairy products and non-dairy snacks on food intake, subjective appetite and cortisol levels in children: a randomized control study. Appl Physiol Nutr Metab. 2021 Sep;46(9):1097-1104. doi: 10.1139/apnm-2020-0909. Epub 2021 Mar 16. PMID 33725464